CLINICAL TRIAL: NCT03381235
Title: The Effects of Exercise on Progression of Disease and Quality of Life in Patients With Retinitis Pigmentosa - a Small Pilot Study
Brief Title: Exercise and RP (AVAMC and Emory)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jiong Yan, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00093690
Record Dates: First submitted 2017-12-13; First posted 2017-12-21 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Retinitis Pigmentosa
Keywords: Exercise; Quality of life; Progression of disease; Retinitis
MeSH Terms: conditions — Retinitis Pigmentosa; Motor Activity; Retinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate exercise (Experimental): Subjects in the moderate exercise group will participate in Spin exercise designed by Dr. Nocera.
  Interventions: Other: Spin exercise
- Mild exercise (No Intervention): Sessions will be focused on balance and stretching.

INTERVENTIONS:
Other: Spin exercise — Each exercise class will consist of 20 minutes of progressive, interval based Spin exercise 2 times a week for 6 months on stationary exercise cycles and will be led by a qualified instructor. The Duration of each session is lengthened based on the progression of the participant and the recommendation of the instructor by 1-2 minutes as needed to a maximum time of 60 minutes per session. Exercise intensity will begin at low levels (50% of maximal heart rate reserve (HRR) and increase by 5% every week (if deemed necessary by the instructor) to a maximum of 75% maximal HRR.
  Arms: Moderate exercise

SUMMARY:
The purpose of this study is to look in humans at the relationship between moderate or little exercise and their potential effects on the retina in patients with Retinitis Pigmentosa (RP).

DETAILED DESCRIPTION:
Human studies have shown that regular exercise may have positive effects on common degenerative diseases such as Alzheimer's disease. Exercise has also shown to improve conditions the eye such as macular degenerations, glaucoma, and cataracts. Mice with retinal degeneration which were exposed to exercise showed that it helped to slow the rate of degeneration. The purpose of this study is to look in humans at the relationship between moderate or little exercise and their potential effects on the retina in patients with Retinitis Pigmentosa (RP).

ELIGIBILITY:
Inclusion Criteria:

* Visual field no less than 10 degrees;
* VA no worse than 20/200 in the better seeing eye.

Exclusion Criteria:

* Not able to tolerate exercise due to an underlying medical condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Brain-Derived Neurotrophic Factor (BDNF) level before and after exercise | Baseline, 3 and 6 months follow up.
  Sertum levels of BDNF in patients before and exercise program will be measured by testing blood

SECONDARY OUTCOMES:
Change in retina vasculature before and after exercise | Baseline, 3 and 6 months follow up.
  Optical Coherence Tomography Angiography (OCTA) will serve as a tool to study retina vasculature, including choroidal, superficial and deep retinal vascular filling status and permeability, before and after exercise.
Change in retinal thickness before and after exercise | Baseline, 3 and 6 months follow up.
  Change in retinal thickness will be evaluated using spectral-domain optical coherence tomography (SD-OCT) before and after exercise.
Change in retinal pigment epithelium (RPE) pigmentation before and after exercise | Baseline, 3 and 6 months follow up.
  Change in retinal RPE pigmentation will be evaluated using Optos wide-field fundus photography before and after exercise.
Change in degrees of vascular attenuation before and after exercise | Baseline, 3 and 6 months follow up.
  Change in degrees of vascular attenuation will be evaluated using Optos wide-field fundus photography before and after exercise.
Change in amount of autofluorescence before and after exercise | Baseline, 3 and 6 months follow up.
  Change in amount of autofluorescence will be evaluated using autofluorescent imaging before and after exercise.
Change in Goldmann Visual Field (GVF) scores | Baseline, 3 and 6 months follow up.
  The final result of a GVF is a diagram "island of vision." The visual field is an island with a central peak and the altitude correlates with the visual sensitivity in a given location.
Change in the National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25) score | Baseline, 3 and 6 months follow up.
  NEI VFQ-25 measures the range of vision-related functioning experienced by persons. The 12 subscales in the NEI VFQ-25 are general vision, near vision, distance vision, driving, peripheral vision, color vision, ocular pain, general health, and vision-specific role difficulties, dependency, social function, and mental health. The subscale scores are calculated by summing the relevant items and transforming the raw scores into a 0 to 100 scale where higher scores indicate better functioning or well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Yan, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Atlanta VA Medical Center, Atlanta, Georgia, United States